CLINICAL TRIAL: NCT02611388
Title: Neurohumor Mechanism of Deferent Frequency Transcutaneous Electrical Acupoint Stimulation(TEAS): A Prospective, Randomized Controlled Trial
Brief Title: Neurohumoral Mechanism of Deferent Frequency Transcutaneous Electrical Acupoint Stimulation(TEAS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: wangqiang (Other)
Responsible Party: Sponsor-Investigator, wangqiang, Doctor, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: XJH-A-2015-10-28
Record Dates: First submitted 2015-11-15; First posted 2015-11-20 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 2/10HZ TEAS pretreatment (Experimental): Patients were given 30min of 2/10HZ TEAS before anesthesia
  Interventions: Device: TEAS (transcutaneous electrical acupoint stimulation)
- 10/50HZ TEAS pretreatment (Experimental): Patients were given 30min of 10/50HZ TEAS before anesthesia
  Interventions: Device: TEAS (transcutaneous electrical acupoint stimulation)
- fake stimulation (Sham Comparator): Patients were only attached electrodes without electric current
  Interventions: Device: fake stimulation

INTERVENTIONS:
Device: TEAS (transcutaneous electrical acupoint stimulation) — 2/10HZ Electric stimulation was given through electrode attached to specific acupoints
  Arms: 2/10HZ TEAS pretreatment
Device: TEAS (transcutaneous electrical acupoint stimulation) — 10/50HZ Electric stimulation was given through electrode attached to specific acupoints
  Arms: 10/50HZ TEAS pretreatment
Device: fake stimulation — Patients were only attached electrodes without electric current
  Arms: fake stimulation

SUMMARY:
The purpose of this study is to explore the neurohumoral mechanism of deferent frequency TEAS pretreatment.

DETAILED DESCRIPTION:
Patients were randomly assigned to three groups, receiving TEAS 30min before anesthesia. The frequency of high frequency group is set to 10/50HZ, low frequency group is 2/10HZ, and the fake stimulation group only attach electrodes without electric current. Acupoint selection is bilateral Neiguan points(PC6). Venous blood is collected 4ml before and immediately after TEAS respectively. Heart rate variability is monitored continuously during the 30min TEAS. The adverse events recorded.

ELIGIBILITY:
Inclusion Criteria:

* Age 18yrs-65yrs
* ASA 1-2
* Scheduled for elective operation under general anesthesia
* BMI 18-30kg/m2
* Informed consented

Exclusion Criteria:

* Contraindications to TEAS
* Communication difficulty with researchers
* Addicted to alcohol, analgesics or other drugs
* Cardiac insufficiency or high blood pressure without controlled
* Hepatic or renal dysfunction
* Participate in the other clinical trial 3 month before the enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-04 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Plasma concentration of epinephrine(ng/L) | change of TEAS 0 and 30 minutes
Plasma concentration of norepinephrine(ng/L) | change of TEAS 0 and 30 minutes

SECONDARY OUTCOMES:
Heart rate variability | During 30min TEAS
plasma concentration of glucocorticoid(μg/L) | change of TEAS 0 and 30 minutes
plasma concentration of aldosterone(ng/L) | change of TEAS 0 and 30 minutes
plasma concentration of renin(ng/L) | change of TEAS 0 and 30 minutes
plasma concentration of β-endorphin(ng/L) | change of TEAS 0 and 30 minutes

REFERENCES:
- [Background] Lu Z, Dong H, Wang Q, Xiong L. Perioperative acupuncture modulation: more than anaesthesia. Br J Anaesth. 2015 Aug;115(2):183-93. doi: 10.1093/bja/aev227. PMID 26170347